CLINICAL TRIAL: NCT01153217
Title: MULTICENTRE STUDY TO ASSESS CHANGES IN BONE MINERAL DENSITY OF THE SWITCH FROM TENOFOVIR TO ABACAVIR IN HIV-1-INFECTED SUBJECTS WITH LOSS OF BONE MINERAL DENSITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Sílvia Gel, Dra. Eugenia Negredo, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSTEOTENOFOVIR
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: HIV
Keywords: Tenofovir; HIV-infection; BMD; Osteoporosis; Osteopenia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Osteoporosis; Bone Diseases, Metabolic | interventions — abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abacavir (Experimental): Switch from tenofovir to abacavir
  Interventions: Drug: Switch from tenofovir to abacavir
- tenofovir (No Intervention): Follow same ART regimen

INTERVENTIONS:
Drug: Switch from tenofovir to abacavir — Switch from tenofovir to abacavir
  Other Names: Abacavir
  Arms: Abacavir

SUMMARY:
Most of studies have not found any consistent drug-specific association with bone loss and controversial data with respect the effect of protease inhibitors (PIs) have been published. The more evident finding with respect to this issue is the more pronounced decrease of bone mineral density (BMD) in patients during the first weeks of receiving a tenofovir (TDF)-containing regimen, probably by the effect of TDF on phosphorus balance and vitamin D metabolism.

DETAILED DESCRIPTION:
The prevalence of osteoporosis in HIV-infected patients could be more than three times greater compared with HIV-uninfected subjects, according to the results of a meta-analytical review of cross-sectional published studies. The analysis includes data from 884 HIV-infected patients and 654 HIV-uninfected controls. Sixty-seven percent of HIV population had reduced bone mineral density (BMD), of whom 15% had osteoporosis (OR of 6.4 and 3.7, respectively, compared with HIV-uninfected controls).

In the same meta-analysis, when authors evaluated the role of antiretroviral therapy (ART) on BMD, comparing 202 antiretroviral-naive with 824 ART-treated patients, patients on treatment had a 2.5-fold increased odds of prevalent reduced BMD and osteoporosis. And finally, when 410 non-protease inhibitor (PI)-treated HIV patients were compared with 791 patients receiving a PI-containing regimen, those on PIs had increased odds of reduced BMD and osteoporosis.

As well, other studies support data of an impaired BMD in HIV-infected patients after starting antiretroviral therapy. These results let us confirm that HIV itself and antiretroviral therapy contribute to decrease the BMD.

However, most of studies have not found any consistent drug-specific association with bone loss and controversial data with respect the effect of PIs have been published. The more evident finding with respect to this issue is the more pronounced decrease of BMD in patients during the first weeks of receiving a tenofovir (TDF)-containing regimen, probably by the effect of TDF on phosphorus balance and vitamin D metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (=/+18 years old) having a diagnosis of HIV-1 infection.
2. Current HAART including tenofovir plus emtricitabine/lamivudine plus a PI, a NNRTI or raltegravir started at least 12 months before.
3. T-score ≤-2 measured by DEXA (within the last 6 months).
4. Maintained undetectable plasma HIV-1 RNA (VL < 50 copies/mL) for at least 12 months.
5. Absence of suspected or documented resistance mutations in the RT associated to abacavir.
6. Voluntary written informed consent.

Exclusion Criteria:

1. History of intolerance, toxicity or virological failure to abacavir.
2. HLA B*5701 positive.
3. Secondary osteoporosis/osteopenia (vitamin D or testosterone deficit, thyroid disease, …)
4. Therapy with biphosphonates within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | From baseline to week 48
t-score change | From baseline to week 48

SECONDARY OUTCOMES:
viral load | Evolution from baseline to week 48
CD4 T lymphocytes count | Evolution from baseline to week 48
Resistance test | If virological failure occurs
Lipid parameters (total, HDL-, LDL-cholesterol and triglyceride levels) | Evolution from baseline to week 48
Adverse Events | From baseline to week 48

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Lluita contra la SIDA Foundation, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona

REFERENCES:
- [Derived] Negredo E, Domingo P, Perez-Alvarez N, Gutierrez M, Mateo G, Puig J, Escrig R, Echeverria P, Bonjoch A, Clotet B. Improvement in bone mineral density after switching from tenofovir to abacavir in HIV-1-infected patients with low bone mineral density: two-centre randomized pilot study (OsteoTDF study). J Antimicrob Chemother. 2014 Dec;69(12):3368-71. doi: 10.1093/jac/dku300. Epub 2014 Aug 13. PMID 25125679